CLINICAL TRIAL: NCT07266610
Title: Effects of Deep Neck Stabilizers Retraining With Pressure Biofeedback on Cervical Pain, Range of Motion and Temporomandibular Dysfunction in Patients With Chronic Neck Pain
Brief Title: Effects of Neck Stabilizers Retraining on Chronic Neck Pain
Acronym: PBU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Umber Nawaz, Assistant Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/024; U1111-1331-6077 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain Musculoskeletal; Chronic Neck Pain
Keywords: Chronic neck pain; Deep neck stabilizers; Pressure biofeedback; Temporomandibular dysfunction
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: 2 groups Experimental group (Group 1): deep neck stabilizers training through pressure biofeedback, along with a traditional exercise program
  Control group (Group 2): traditional exercise program
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Biofeedback-assisted deep neck flexor retraining ) (Experimental): Each session includes TENS and hot pack therapy, crook lying exercises with a 20 mmHg pressure biofeedback sensor, the Cranio-Cervical Flexion Test, and neck and shoulder stretches. Data will be collected at the initial point, after 3 weeks, and once more at the 6-week point.
  Interventions: Other: Biofeedback-assisted deep neck flexor retraining
- Group 2 (Conventional exercises) (Active Comparator): Each session begins with TENS and hot pack therapy, followed by stretching and strengthening exercises for neck and shoulder muscles. Data will be collected at the initial point, after 3 weeks, and once more at the 6-week point.
  Interventions: Other: Conventional exercises

INTERVENTIONS:
Other: Biofeedback-assisted deep neck flexor retraining — The experimental group will receive deep neck stabilizer training with pressure biofeedback and traditional exercises for six weeks, three times weekly.
  Arms: Group 1 (Biofeedback-assisted deep neck flexor retraining )
Other: Conventional exercises — The control group will engage in a traditional exercise program for 6 weeks, meeting three times weekly
  Arms: Group 2 (Conventional exercises)

SUMMARY:
The present study aims to evaluate the effects of deep neck stabilizers retraining with pressure biofeedback on cervical range of motion, pain, and temporomandibular dysfunction in patients with chronic neck pain.

Participants will receive biofeedback-assisted deep neck flexor retraining in one group, while the other group will perform conventional exercises. The neurological connection between the TMJ and neck means that therapies such as neck flexion exercises and biofeedback can alleviate neck pain and jaw issues.

DETAILED DESCRIPTION:
Chronic neck pain is increasingly affecting young adults in Pakistan. This rise is linked to poor posture, being overweight, aging, and various other factors. Weakness in deep neck muscles can affect neck stability. The craniocervical flexion test (CCFT) is useful for evaluating and engaging these muscles. The jaw joint (Temporomandibular joint) and the neck are closely connected through shared nerves. Therefore, problems in the neck can lead to jaw issues (pain and difficulty moving the jaw). Using biofeedback to train deep neck muscles helps improve muscle control, posture, and reduces stress on surface and jaw muscles, easing TMJ symptoms. However, many studies on deep neck stabilizer (DNS) exercises don't focus on jaw problems. This study utilizes pressure biofeedback to relieve pain, improve mobility, and reduce jaw tension by promoting better neck posture.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Chronic neck pain (duration more than 3 months and less than 1 year and 6 months)
* TMJ Dysfunction (RCD TMJ Axis I Confirmation on Helkino Index) Fonseca Anamnestic Index (FAI) 20-65 score mild to moderate

Exclusion Criteria:

* Traumatic neck injury
* Neurological disorders
* Cervical spine infection or surgery
* Cancer

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Temporomandibular dysfunction | 6 weeks
  Mandibular Functional Impairment Questionnaire
Pain Intensity | 6 weeks
  Numeric Pain Rating Scale will be used
Cervical Range of Motion | 6 weeks
  Inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Society for the Rehabilitation of the Disabled (PSRD), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sikka I, Chawla C, Seth S, Alghadir AH, Khan M. Effects of Deep Cervical Flexor Training on Forward Head Posture, Neck Pain, and Functional Status in Adolescents Using Computer Regularly. Biomed Res Int. 2020 Oct 5;2020:8327565. doi: 10.1155/2020/8327565. eCollection 2020. PMID 33083487
- [Result] Alagingi NK. Chronic neck pain and postural rehabilitation: A literature review. J Bodyw Mov Ther. 2022 Oct;32:201-206. doi: 10.1016/j.jbmt.2022.04.017. Epub 2022 Apr 20. PMID 36180150
- [Result] Aguiar ADS, Nogueira Carrer HC, de Lira MR, Martins Silva GZ, Chaves TC. Patient-Reported Outcome Measurements in Temporomandibular Disorders and Headaches: Summary of Measurement Properties and Applicability. J Clin Med. 2021 Aug 26;10(17):3823. doi: 10.3390/jcm10173823. PMID 34501273
- [Result] Craciun MD, Geman O, Leuciuc FV, Holubiac IS, Gheorghita D, Filip F. Effectiveness of Physiotherapy in the Treatment of Temporomandibular Joint Dysfunction and the Relationship with Cervical Spine. Biomedicines. 2022 Nov 17;10(11):2962. doi: 10.3390/biomedicines10112962. PMID 36428529